CLINICAL TRIAL: NCT02630329
Title: Adnexectomy for Benign Gynaecological Pathology by Natural Orifice Transluminal Endoscopy or Laparoscopy
Brief Title: Notes Adnexectomy for Benign Pathology Compared to Laparoscopic Excision
Acronym: NOTABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imelda Hospital, Bonheiden (Other)
Responsible Party: Principal Investigator, Dr Jan Baekelandt, MD, Dr, Imelda Hospital, Bonheiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B689201526268
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Natural Orifice Endoscopic Surgery; Disease, Adnexal; Laparoscopic Surgery
Keywords: NOTES; Benign adnexal disease; Laparoscopy
MeSH Terms: conditions — Adnexal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vNOTES adnexectomy (Experimental): Vaginal Natural Orifice Transluminal Endoscopic Surgery
  Interventions: Procedure: vNOTES adnexectomy
- LSC adnexectomy (Active Comparator): Laparoscopic adnexectomy
  Interventions: Procedure: Laparoscopic adnexectomy

INTERVENTIONS:
Procedure: vNOTES adnexectomy — Surgical removal of one or both adnexa by a natural orifice transluminal endoscopic surgical technique using a colpotomy (transvaginal incision)
  Arms: vNOTES adnexectomy
Procedure: Laparoscopic adnexectomy — Surgical removal of one or both adnexa by transabdominal laparoscopy
  Arms: LSC adnexectomy

SUMMARY:
Objective: To compare vNOTES (vaginal Natural Orifice Transluminal Endoscopic Surgery) and established laparoscopic removal of benign adnexal masses Study design: Randomized controlled/single center/single-blinded/parallel-group/non-inferiority/efficacy trial.

Study population: Women aged 18 to 70 years with symptomatic or persistent benign adnexal masses detected by clinical examination and ultrasound.

Randomization: Women will be randomly allocated to undergo one of two techniques for removal of the benign adnexal mass immediately before surgery by using a computer generated randomization list. The investigators will use stratified randomization according to the cyst diameter.

Intervention: Women will be treated by a surgeon who is not blinded to the treatment allocation and who is equally skilled in performing both techniques. In the intervention group a vNOTES technique will be used.

Control: In the control group surgery will be done by a classical laparoscopic technique.

Participants, nursing staff and outcome assessors will be blinded.

Main study parameters/endpoints:

Primary outcomes: successful removal of a benign adnexal mass without spill. Secondary outcomes: the proportion of women discharged the same day based on their own preference; postoperative pain scores using a VAS (Visual Analogue Scale) measured between day 1 till 7 by the participating women following surgery and the total amount of analgesics used as described in the standardized pain treatment protocol between day 1 till 7; postoperative infection defined by lower abdominal pain with fever > 38°C and positive clinical signs or laboratory findings; per- or postoperative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery; duration of the surgical procedure; incidence and intensity of dyspareunia recorded by the participants at 3 and 6 months by self-reporting using a simple questionnaire and VAS scale; sexual wellbeing recorded by the participants at 3 and 6 months by SSFS (Short Sexual Functioning Scale); direct costs associated up to 6 weeks after the surgical intervention with both procedures.

DETAILED DESCRIPTION:
1. Objectives of the NOTABLE Trial

The primary research questions of this IDEAL stage 2b efficacy trial are as follows: is a vNOTES adnexectomy at least as effective compared to the standard transabdominal laparoscopic approach (LSC) for removing a benign adnexal mass without spill? (non-inferiority design)

Secondary research questions are:

* Do more women treated by vNOTES prefer to leave the hospital on the day of surgery compared to LSC?
* Do women treated by vNOTES suffer from less pain compared to women treated by LSC in the first postoperative week?
* Is the removal of a benign adnexal mass by vNOTES faster compared to LSC?
* Does a vNOTES cause more pelvic infection or other complications compared to LSC?
* Does a vNOTES cause more hospital readmissions within 6 weeks following surgery compared to LSC?
* Does a vNOTES approach result in more women reporting dyspareunia, less sexual wellbeing or less health-related quality of life at 3 or 6 months after surgery when compared to women treated by LSC?
* What are the direct and indirect costs up to 6 weeks of a vNOTES compared to LSC?

TRIAL DESIGN 2.1. Design A single center, single-blinded, parallel group randomized, non-inferiority efficacy trial.

2.2. Simple pilot randomized trial: minimal extra workload 2.3. Time schedule Based upon the mean number of laparoscopic adnexectomies performed annually at the department of Obstetrics and Gynecology of the participating center (36) the investigators estimate that the duration of recruitment will be 21 months. Based upon the follow up (6 months) and the period of analysis/reporting (3 months) the total study period will be 2.5 years.

2.4. Participating center Department of Obstetrics and Gynecology Imeldahospital Imeldalaan 9 2820 Bonheiden Belgium

3. ELIGIBILITY, CONSENT AND RANDOMIZATION 3.1. Screening and consent prior to surgery All women aged 18 to 70 years regardless of parity presenting with a symptomatic or asymptomatic persistent benign adnexal mass on clinical examination confirmed by ultrasound are eligible for inclusion. The diagnosis of benign adnexal mass will be based upon the prospectively validated IOTA classification(International Ovarian Tumour Analysis Group) simple ultrasound rules to distinguish between benign and malignant adnexal masses.

3.2. Determining eligibility All women aged 18 to 70 years regardless of parity presenting with a symptomatic or asymptomatic persistent benign adnexal mass on clinical examination who provide consent to participation are eligible in the NOTABLE trial based on the findings of the ultrasound findings and will be randomized before the procedure.

3.3. Randomization If the woman is eligible for the NOTABLE trial, the trial secretary will obtain a randomized allocation the day before surgery. This will be done using a randomization list generated by a free computer software program offered by Research Randomizer (https://www.randomizer.org). The random sequence generation will be concealed using sequentially numbered opaque sealed envelopes. The envelope will be opened by the nurse assistant on the day before the surgical intervention for logistic reasons. The investigators will use stratified randomization in this small pilot RCT (randomized controlled trial) according to the cyst diameter.

3.4. Patients with strong preference for treatment A minority of women will express a clear preference for one of both treatments (e.g. strong desire to have no scar) and for this reason will not wish to be randomized between surgical treatments. To investigate how outcomes vary by choice, these women could be followed up in exactly the same way as for those women randomized into the NOTABLE trial. A formal non-randomized follow-up of these women will not be done for simple logistical reasons.

3.5. Stratification of randomization A blocked randomization procedure will be used to avoid chance imbalances for the parameter 'cyst diameter'.

To avoid any possibility of foreknowledge, the randomized allocation will not be given until all eligibility and stratification data have been given.

4. TREATMENT ALLOCATIONS 4.1. Surgical procedures The principal investigator, who has training and experience in both laparoscopy and NOTES, will perform all surgical procedures. He is therefore not blinded. All vNOTES participants will be blinded by three superficial "mock" skin incisions similar to those routinely done with the laparoscopic technique.

4.1.1 vNOTES adnexectomy This is the surgical procedure done in the intervention arm of the NOTABLE trial.

4.1.2 LSC adnexectomy This is the surgical procedure done in the control arm of the NOTABLE trial. 5. FOLLOW-UP AND OUTCOME MEASURES 5.1. Clinical assessments 5.1.1 Format PROMs will be collected using a postal questionnaire, which will include a combination of disease specific and generic measurement instruments.

The postal questionnaires will be sent from the NOTABLE Trial Office with postage paid envelopes two weeks before the due date. Reminders will be sent to the participants if the questionnaire is not returned within one week of the due date and attempts will be made to contact the women by phone if the questionnaire is not returned by two weeks after the due date.

5.1.2 Timing of assessments The primary outcome will be measured clinically at the end of the surgical procedure. In addition patient reported outcome measures (PROMs) will take place the evening of the surgical intervention (return home), during the first postoperative week (pain by Visual Analogue (VAS)scores and analgetic drugs) and at 3 and 6 months (dyspareunia/ sexual well being/ health related quality of life). Clinical physician assessment will take place the evening of the surgical intervention (return home) and during the first six weeks following surgery (pelvic infection, surgical complications, hospital readmission rate).

5.2. Primary clinical outcome measure The proportion of women successfully treated by removing the adnexal mass without spill, using a dichotomous outcome measure, will be used as a measure of efficacy.

5.3. Secondary clinical outcome measures

The following secondary outcomes will be measured:

* The proportion of women admitted in-hospital for at least one night observation based on their own preference, as a dichotomous outcome.
* Postoperative pain scores, as an ordinal outcome, measured using a Visual Analogue Scale (VAS) scale twice daily from day 1 till 7 self-reported by the participating women. VAS scores range from 0=no pain to 10= worst imaginable pain.
* Postoperative pain defined by the total amount of analgesics used as described in the standardized pain treatment protocol, as a continuous outcome.
* Postoperative infection as a dichotomous outcome.
* Per- or postoperative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery, as a dichotomous outcome.
* Hospital readmission within 6 weeks following surgery, as a dichotomous outcome.
* Incidence and intensity of dyspareunia recorded by the participants at 3 and 6 months by self-reporting using a simple questionnaire and Visual Analogue Scale (VAS) scale, as a dichotomous and ordinal outcome. VAS scores range from 0=no pain to 10= worst imaginable pain.
* Sexual wellbeing at baseline, at 3 and 6 months by self-reporting the Short Sexual Functioning Scale (SSFS). The SSFS is a questionnaire with 7 open ended questions on sexual wellbeing.
* Health-related quality of life, at baseline, at 3 and 6 months by self-reporting the EQ-5D-3L tool consisting of a questionnaire on 5 domains and a scale ranging from 0=worst possible health-related quality of life to 100 = best possible health-related quality of life.
* Duration of surgery measured as the time in minutes from the insertion of the bladder catheter to the end of vaginal/abdominal wound closure, as a continuous outcome.

5.4. Health economic outcomes The direct and indirect costs of both techniques up to 6 weeks after the surgical intervention will be calculated.

6. ACCRUAL AND ANALYSIS 6.1. Sample size The sample size for this trial has been chosen to give good statistical power to preclude any clinically important inferiority of vNOTES compared to laparoscopy and is based on evidence retrieved from a systematic review of the literature and a RCT comparing the excision of mature teratoma using culdotomy with and without laparoscopy. Based on the power calculations for the primary outcome and two secondary outcomes and assuming a loss-to-follow-up rate of 10% the investigators decided to include 66 study participants in the NOTABLE trial.

6.2. Projected accrual and attrition rates It is anticipated that recruitment of participants will take two years. Based upon the mean number of laparoscopic adnexectomies performed annually at the department of Obstetrics and Gynecology of the participating center (36) the investigators estimate that the duration of recruitment will be 21 months. Based upon the follow up (6 months) and the period of analysis/reporting (3 months) the total study period will be 2.5 years. First publication will be possible within four years of trial commencement.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18 to 70 years regardless of parity with a symptomatic adnexal mass presumed to be benign based on ultrasound examination by applying the IOTA simple rules
* All women aged 18 to 70 years regardless of parity with an asymptomatic persistent adnexal mass presumed to be benign based on ultrasound examination by applying the IOTA simple rules
* Written informed consent obtained prior to surgery

Exclusion Criteria:

* History of hysterectomy by any technique
* History of rectal surgery
* Suspected rectovaginal endometriosis
* Suspected endometriotic cyst
* Solid adnexal mass
* High suspicion of adnexal malignancy based on clinical, ultrasound or biochemical findings
* History of pelvic inflammatory disease, especially prior tubo-ovarian or pouch of Douglas abscess
* Active lower genital tract infection e.g. Chlamydia, N. gonorrhoeae
* Virgo
* Pregnancy
* Need for other uterine surgical intervention (i.e. endometrial ablation, resection, myomectomy or hysterectomy)
* Additional pathology necessitating hysterectomy
* Failure to provide written informed consent prior to surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-02-03 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Successful removal of adnexal mass without spill | Intraoperative
  The proportion of women successfully treated by removing the adnexal mass without spill, using a dichotomous outcome measure, will be used as a measure of efficacy.

SECONDARY OUTCOMES:
Discharge from the hospital the day of the surgical intervention | Dichotomous outcome measured on the day of the surgical intervention
  The proportion of women discharged the same day based on their own preference, as a dichotomous outcome. The decision to discharge or to admit to hospital for the night will be based solely on the choice of the woman to return home the same day or stay overnight.
Postoperative pain scores | The first week after the surgical intervention
  Postoperative pain scores, as an ordinal outcome, measured using a VAS scale twice daily from day 1 till 7 self-reported by the participating women
The use of analgesics for postoperative pain | The first week after the surgical intervention
  Postoperative pain defined by the total amount of analgesics used as described in the standardized pain treatment protocol, as a continuous outcome.
Postoperative infection | The first six weeks after the surgical intervention
  Postoperative infection defined by lower abdominal pain with fever > 38°C and positive clinical signs or laboratory findings, detected during the first six weeks of surgery, as a dichotomous outcome.
Complications | The first six weeks after the surgical intervention
  Per- or postoperative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery, as a dichotomous outcome
Hospital readmission | The first six weeks after the surgical intervention
  The proportion of women readmitted to hospital within six weeks of surgery, as a dichotomous outcome
Pain during sexual intercourse | At baseline, 3 months and 6 months after the surgical intervention
  Incidence and intensity of dyspareunia recorded by the participants at 3 and 6 months by self-reporting using a simple questionnaire and VAS scale, as a dichotomous and ordinal outcome
Sexual well being | At baseline, 3 months and 6 months after the surgical intervention
  Sexual wellbeing at baseline, at 3 and 6 months by self-reporting using the SSFS (Short Sexual Function Scale).
Duration of the surgical intervention | Intraoperative
  Duration of surgery measured as the time in minutes from the insertion of the bladder catheter to the end of vaginal/abdominal wound closure, as a continuous outcome
Direct and indirect costs | Up to 6 weeks postoperative
  Calculating the comparative direct costs of both techniques up to 6 weeks after the surgical intervention
Health-related quality of life | At baseline, at 3 months and 6 months after the surgical intervention
  Health-related quality of life, at baseline, at 3 and 6 months by self-reporting the EQ-5D-3L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jan Baekelandt, MD, Principal Investigator — Imelda Hospital, Bonheiden
Locations (1):
- Imelda Hospital, Bonheiden, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Interim analyses of major endpoints will be supplied, in strict confidence, to an independent Data Monitoring and Ethics Committee (DMEC) along with updates on results of other related studies, and any other analyses that the DMEC may request.

REFERENCES:
- [Background] Wang PH, Lee WL, Juang CM, Tsai WY, Chao HT, Yuan CC. Excision of mature teratoma using culdotomy, with and without laparoscopy: a prospective randomised trial. BJOG. 2001 Jan;108(1):91-4. doi: 10.1111/j.1471-0528.2001.00003.x. PMID 11213011
- [Result] Baekelandt J. Poor man's NOTES: can it be a good approach for adhesiolysis? A first case report with video demonstration. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):319. doi: 10.1016/j.jmig.2014.11.001. Epub 2014 Nov 10. PMID 25460516
- [Result] Yang YS, Hur MH, Oh KY, Kim SY. Transvaginal natural orifice transluminal endoscopic surgery for adnexal masses. J Obstet Gynaecol Res. 2013 Dec;39(12):1604-9. doi: 10.1111/jog.12108. Epub 2013 Jul 22. PMID 23875997
- [Result] Ghezzi F, Cromi A, Uccella S, Bogani G, Serati M, Bolis P. Transumbilical versus transvaginal retrieval of surgical specimens at laparoscopy: a randomized trial. Am J Obstet Gynecol. 2012 Aug;207(2):112.e1-6. doi: 10.1016/j.ajog.2012.05.016. Epub 2012 May 23. PMID 22704765
- [Result] Medeiros LR, Rosa DD, Bozzetti MC, Fachel JM, Furness S, Garry R, Rosa MI, Stein AT. Laparoscopy versus laparotomy for benign ovarian tumour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD004751. doi: 10.1002/14651858.CD004751.pub3. PMID 19370607
- [Derived] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BWJ, Bosteels JJA. Transvaginal natural orifice transluminal endoscopic surgery (vNOTES) adnexectomy for benign pathology compared with laparoscopic excision (NOTABLE): a protocol for a randomised controlled trial. BMJ Open. 2018 Jan 10;8(1):e018059. doi: 10.1136/bmjopen-2017-018059. PMID 29326183

DOCUMENTS (1):
  • Study Protocol (2015-12-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02630329/Prot_000.pdf